CLINICAL TRIAL: NCT04958837
Title: Effects of FIFA 11+ With and Without Dynamic Core Stability Training on Balance and Dynamic Knee Valgus in Amateur Soccer Players at Risk of Anterior Cruciate Ligament Injury
Brief Title: Effects of FIFA 11+ With Dynamic Core Stability Training on Balance and Dynamic Knee Valgus in Amateur Soccer Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/1105
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Injury Prevention; Postural Balance
Keywords: Exercise training; knee joint; soccer

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to Interventional Group A (FIFA 11+ with dynamic core stability training protocol) or Interventional Group B/ Control Group (FIFA 11+ protocol) for the whole duration of the study.
Who Masked: Participant
Masking Description: It will be a single blinded study. Only the participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ with dynamic core stability training (Experimental): Participants in this group will undergo FIFA 11+ protocol along with additional Core training exercises including leg raises, crunches, superman, plank hip twist, and supine bridge will be given. Each exercise plan will be progressively increased.
  Interventions: Other: FIFA 11+ protocol with additional Core training exercises
- FIFA 11+ protocol (Active Comparator): Participants in this group will undergo traditional FIFA 11+ protocol which consists of slow paced running exercises, strength, plyometric & Balance exercises and high speed running with planting/cutting
  Interventions: Other: FIFA 11+ protocol

INTERVENTIONS:
Other: FIFA 11+ protocol with additional Core training exercises — Slow paced running exercises of 8 minutes' duration (2 rounds each), followed by Strength, plyometric and balance exercises including 3 sets of 20-30 sec of The Bench, Sideways Bench each side, Nordic Hamstring strengthening, single leg stance balance training, squatting and high speed running. The protocol will end with additional core training exercises including leg raises, crunches, superman, plank hip twist, and supine bridge. Each exercise plan will be progressively increased. Core training will be followed by 30 sec stretch of major muscle groups.
  Arms: FIFA 11+ with dynamic core stability training
Other: FIFA 11+ protocol — Slow paced running exercises of 8 minutes' duration including running straight, running with hip out, running hip in, running circling partner, running shoulder contact and running quickly forward and backwards (2 rounds each), followed by Strength, plyometric and balance exercises including The Bench, Sideways Bench each side, Nordic Hamstring strengthening and single leg stance balance training, squatting and jumping. All exercises will be progressively increased as per established protocol. The final phase of the study includes fast running for 2 minutes.
  Arms: FIFA 11+ protocol

SUMMARY:
The incidence of soccer-related injuries is reported to have the highest rate amongst all sports. To reduce the incidence of soccer injuries in youth and amateur soccer players, an injury prevention framework namely FIFA 11+ was established. Although the FIFA 11+ is a comprehensive warm-up and training program for soccer players, yet in the second component focusing on strength and plyometric training, the exercises consist of only static core training whereas dynamic core training is not included in the protocol. Hence this study will observe the effect of including dynamic core training targeting the remaining core musculature as well in the FIFA 11 + program for risk factor modification and correction of muscular imbalance.

DETAILED DESCRIPTION:
Soccer (football) is one of the most popular sports in the world. Intense soccer actions (i.e., acceleration, decelerations, change of direction, sprinting, tackling, running, being tackled, and shooting, twisting, turning, jumping and landing during the game) in addition to high impact and forceful body contacts during practice sessions and matches predispose the athletes to injuries. various contributing factors of these injuries include muscular imbalance, joint instability, lack of proper training and inadequate rehabilitation. Poor landing mechanics, specifically, increased dynamic knee valgus, is also associated with increased risk for lower limb injury, particularly ACL injury. The modifiable factors are shown to be responsive to different types of trainings. In fact neuromuscular factors are involved in control of dynamic knee stability, hamstrings and quadriceps imbalances, asymmetry of legs and core dysfunction. The latest FIFA 11+ developed in 2006 was designed to be used as pre-training protocol to improve the components of physical fitness that might contribute to injury prevention. In this program, there is a combination of three major exercise regime components: an initial running and stretching exercises, second component of strength, plyometric and balance exercises, ending with high speed planting and cutting exercises. One of the component of this program involves the training of core musculature. While the core muscles (including muscles of trunk and pelvis) do not cross the knee joint, yet core stability can modulate the lower limb alignment and loading during dynamic tasks. Hence, this study will be conducted to find whether there is any effect of including dynamic core training in the FIFA 11+ program in order to correct muscular imbalances and ultimately risk factor modification. A two-arm single blinded randomized controlled trial will be conducted to find out the dynamic knee valgus alignment, postural stability and single leg athletic stability and lower limb muscles strength, while the secondary outcomes would include lung function tests (FEV1, FVC & FEV1/FVC ratio). In the control group, standard FIFA 11+Protocol will be followed consisting of slow paced running exercises followed by strength, plyometric and balance training. In the experimental group, FIFA 11+ protocol along with additional dynamic core exercises will be followed including leg raises, crunches, superman, plank hip twist, and supine bridge.All exercises in both groups will be progressively increased as per established protocol. Training will be provided 3-4 Times a week for 8 Weeks on alternate days.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females
2. Between the Age of 13-25 Years
3. Participants will be selectively recruited with high risk of ACL/Knee Injury.
4. Individuals of selected football academies, performing routine exercise according to the football academy.
5. Able to provide informed consent by them self or from guardians

Exclusion Criteria:

1. Players having history of any Musculoskeletal Disorder or injury
2. Players having recent injury resulting in at least 10-30 days off time from full training or matches.
3. Players having history of skeletal trauma such as lower limb fractures.
4. Players having history of any severe medical problems hindering regular participation in evaluation or training.
5. Players using any nutritional supplements.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic Knee Valgus | 8 weeks
  Dynamic knee valgus will be measured using Motion Analysis System and expressed in form of degrees.
Single Leg Athletic Stability | 8 weeks
  Single Leg Athletic Stability will be measured using objective balance evaluation system.

SECONDARY OUTCOMES:
Lung function Test | 8 weeks
  FEV1 & FCV will be measured using hand held spirometer dynamometer and expressed in form Liters.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Foundaion University Institute of Rehabilitation Sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No